CLINICAL TRIAL: NCT05079035
Title: A Phase 2, 52-Week Trial of TTAX03 vs. Saline as a Single Intra-articular Injection in Kellgren-Lawrence Grade 3-4 Knee OA
Brief Title: Lyophilized and Micronized Particulate Human Amniotic and Umbilical Cord (TTAX03) for KL Grade 3-4 Knee OA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioTissue Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTAX03-CR005
Record Dates: First submitted 2021-09-22; First posted 2021-10-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: TTAX03 (Experimental): TTAX03 is a sterile, lyophilized and micronized particulate human AM and UC product manufactured using aseptic processing followed by terminal sterilization by gamma irradiation in compliance with current Good Tissue Practices (cGTP) and current Good Manufacturing Practices (cGMP) to preserve extracellular matrices and growth factors/cytokines therein without any living cells. TTAX03 is suspended in a volume of 2.0mL of sterile, preservative free 0.9% NaCl.
  Interventions: Biological: TTAX03
- Control: Saline (Placebo Comparator): 2.0mL of sterile, preservative free 0.9% NaCl alone
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: TTAX03 — Lyophilized and Micronized Particulate Human Amniotic and Umbilical Cord
  Arms: Experimental: TTAX03
Biological: Saline — 2 mL Sterile, preservative free 0.9% NaCl
  Arms: Control: Saline

SUMMARY:
It is hypothesized that a single Intra-articular Injection of TTAX03, 100mg in 2mL of saline, will have more benefit with respect to the proportion of responders 12 weeks post-injection than an equal volume of saline, based on the OMERACT-OARSI responder criteria.

DETAILED DESCRIPTION:
This trial is designed as a Phase 2 randomized, placebo controlled, double-blinded parallel design to be conducted at multiple sites throughout North America. One dose level of TTAX03 (100 mg) will be tested against an equal volume of saline, which is the suspension vehicle (i.e., excipient). Each subject will receive a single IA injection into the knee under local anesthesia, with two safety follow-up visits in the first eight days and a third at the end of two weeks post injection. Subsequent visits will occur at the end of 6 and 12 weeks for evaluation of response, with the end of 12 weeks being the primary endpoint. Additional visits will occur at 6, 9 and 12 months (end of weeks 26, 39, 52) to evaluate duration of benefit and overall impression of change from baseline, as well as safety. The primary endpoint will be assessed at 12 weeks post receiving the assigned Intra-articular injection.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* ≥ 35 and ≤ 85 years of age (until a cap of 30 subjects < 50 years of age is reached, at which point this will convert to ≥ 50 and ≤ 85 years of age)
* Able to reliably complete the KOOS self-administered questionnaire
* Clinical diagnosis of OA of the index knee, with pain onset more than one year prior to screening according to subject recall
* KL grade 3 or 4 in the index knee
* Pain score (KOOS) over the past week ≥ 70 in the index knee at Screening (the index knee will be the more painful knee by ≥ 20 in the case of bilateral disease)
* A ≥ 3 months history of insufficient pain relief from IA hyaluronic acid or a ≥ 3 months history of insufficient pain relief from IA corticosteroids, unless they are medically contraindicated for the subject
* A ≥ 3 months history of insufficient pain relief from other currently recommended treatments, including weight loss and physical therapy
* Any two of the following:

  * Severe knee pain or stiffness that limits everyday activities, including walking, climbing stairs, and getting in and out of chairs. Finding it hard to walk more than a few blocks without significant pain and need to use a cane or walker
  * Moderate or severe knee pain while resting, either day or night
  * Chronic knee inflammation and swelling that does not improve with rest or medications
* BMI ≤ 40 kg/m2
* Adequate bone marrow function (ANC > 1000 × 109 /L, platelets ≥ 100,000 × 109 /L, Hgb ≥ 10 g/dL)
* Adequate hepatic function (AST/ALT ≤ 1.5 × ULN, total bilirubin ≤ 1.2 × ULN)
* Adequate renal function (creatinine ≤ 1.2 × ULN)
* Negative urine test for opioids (including synthetic opioids)
* If female and of child-bearing potential, willingness to use effective birth control during the study.

Exclusion Criteria:

* Cognitive impairment, mental illness, neuroses or untreated depression that would preclude understanding or reliably completing the patient reported outcome measures
* Non-ambulatory, bedridden, or with active fibromyalgia, radiculopathy, painful peripheral neuropathy, vascular insufficiency, hip OA or other joint disease severe enough to prevent assessment of knee pain or causing functional impairment
* Current use of opioid analgesics, or positive urine laboratory test for opiates during the screening period
* Hyaluronic acid, corticosteroid, platelet rich plasma or stem cells IA knee injections within the prior 3 months, oral or intramuscular corticosteroids within the prior 2 months
* Scheduled knee arthroscopy or knee surgery in either knee within 12 weeks from enrollment
* Known or suspected joint infection of either knee
* History of knee ligament surgery in the past 12 months
* Acute injury to the knee in the past 3 months resulting in difficulty walking for more than 24 hours
* History of inflammatory joint diseases, crystalline diseases such as gout or pseudogout, systemic lupus, rheumatoid arthritis, autoimmune disease or Crohn's disease
* Previous repair of a cruciate ligament, osteochondral autograft transfer, mosaicplasty, subchondral surgery (subchondroplasty) or previously diagnosed subchondral insufficiency fracture
* Comorbid conditions that include the following: known other causes of arthritis (infectious arthritis, or psoriatic arthritis), osteomyelitis, cardiopulmonary disease that limits walking more than knee pain, bone metastases or Paget's disease involving the lower extremities.
* Psoriasis or other acute or chronic inflammatory conditions or infection affecting the skin over the index knee
* Symptoms of locking, intermittent block to range of motion or loose body sensation which could indicate meniscal displacement or an intraarticular loose body in the index knee
* Use of anticoagulants (except for ≤ 81 mg of aspirin per day) or a history of any coagulopathy or bleeding disorder, sickle cell disease
* History of substance abuse in the past 2 years
* Prior or current use of systemic immunosuppressive medications (other than corticosteroids for arthritis), chemotherapy, or history of organ transplant (kidney, heart, lung)
* Prior radiation therapy to the index knee
* Prior treatment with CLARIX FLO, NEOX FLO, or injectable birth tissue products for any indication
* Concurrent treatment, or treatment in the past 90 days, with any investigational agent
* Severe concurrent illness which, in the view of the investigator, would interfere with this 52 week study
* Any condition which, in the opinion of the investigator, would make a patient a poor candidate for this study
* Positive blood pregnancy test or known pregnancy

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Pain Relief and/or Functional Improvement | 12-weeks post Intra-articular Injection
  Proportion of subjects who, at the end of 12 weeks, report improvement from baseline in pain or in function > or = 50% and absolute change > or = 20;
  - or -
  Improvement in at least 2 of the 3 following:
  * pain > or = 20% and absolute change > or = 10
  * function > or = 20% and absolute change > or = 10
  * global assessment > or = 20% and absolute change > or = 10

SECONDARY OUTCOMES:
KOOS Knee Symptoms Subscale | 6,12, 26, 39 & 52 weeks from Baseline versus Saline
  Change from Baseline as a result of the intervention on joint symptoms
KOOS Knee Pain Subscale | 6,12, 26, 39 & 52 weeks from Baseline versus Saline
  Change from Baseline as a result of the intervention on Knee Pain
KOOS Physical Function Subscale | 6,12, 26, 39 & 52 weeks from Baseline versus Saline
  Change from Baseline as a result of the intervention on Physical Function
KOOS Sports and Recreation Subscale | 6,12, 26, 39 & 52 weeks from Baseline versus Saline
  Change from Baseline as a result of the intervention on Sports and Recreation activities
KOOS Quality of Life Subscale | 6,12, 26, 39 & 52 weeks from Baseline versus Saline
  Change from Baseline as a result of the intervention on joint-specific Quality of Life
Patient Global Impression of Change Questionnaire | 12, 26, 39 & 52 weeks from Baseline versus Saline
  Change from Baseline as a result of the intervention on patient reported Global Impression of Change
Overall Change in Pain Relief Medication Use from Baseline | Over the 52 weeks from Baseline versus Saline
  Change in time to and frequency of use of pain relief medications and intra-articular injection of steroids and/or HA

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - UAB Orthopaedic Surgery, Birmingham, Alabama
  - Alabama Orthopaedic Center, Birmingham, Alabama
  - Tuscon Orthopedic Institute, Tucson, Arizona
  - Horizon Clinical Research, La Mesa, California
  - Gulfcoast Research Institute, Sarasota, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Paragon Sports Medicine, Atlanta, Georgia
  - Ochsner Health Center, Jefferson, Louisiana
  - Manage Sites/The Ohio State University Wexner Medical Center, Sports Medicine The Ohio State University Wexner Medical Center, Sports Medicine, Columbus, Ohio
  - Rothman Orthopaedic Institute, Media, Pennsylvania

IPD SHARING:
Plan to Share IPD: No